CLINICAL TRIAL: NCT00959270
Title: Pennington Center Longitudinal (PCLS)
Brief Title: Pennington Center Longitudinal Study (PCLS)
Acronym: PCLS
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Princiapal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 28027
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Health Behaviors; Development of Health Problems
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a cohort of volunteers that can be studied and followed up into the future for changes in health behaviors and development of health problems.

DETAILED DESCRIPTION:
The PCLS represents an effort to utilize the data collected over the last twenty years during the clinical research studies conducted at Pennington Biomedical Research Center. A cohort will be developed and used for cross-sectional analyses, as well as followed prospectively for the development of a variety of health-related outcomes. Several data sources from the PBRC clinical database will be used to establish the PCLS database, including screening, archive and study-specific data. The only protocol specific to the PCLS study is the collection of blood sample for risk factor determination and storage in the PBRC archive bank, only to be invoked in cases where studies do not include a blood draw as part of their protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* volunteer to Participate

Exclusion Criteria:

* younger than 18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2009-05; Primary Completion 2050-02 (Estimated); Study Completion 2050-02 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional analyses database | twenty-years
  The only protocol specific to the PCLS study is the collection of blood sample for risk factor determination and storage in the PBRC archive bank, only to be invoked in cases where studies do not include a blood draw as part of their protocol. The PCLS represents an effort to utilize a data collection over the last twenty years during the clinical research studies for cross-sectional analyses, as well as followed prospectively for the development of a variety of health-related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Katzmarzyk, PhD, Principal Investigator — Associate Executive director for Population Science
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Camhi SM, Katzmarzyk PT. Differences in body composition between metabolically healthy obese and metabolically abnormal obese adults. Int J Obes (Lond). 2014 Aug;38(8):1142-5. doi: 10.1038/ijo.2013.208. Epub 2013 Nov 12. PMID 24216712
- [Result] Katzmarzyk PT, Greenway FL, Heymsfield SB, Bouchard C. Clinical utility and reproducibility of visceral adipose tissue measurements derived from dual-energy X-ray absorptiometry in White and African American adults. Obesity (Silver Spring). 2013 Nov;21(11):2221-4. doi: 10.1002/oby.20519. Epub 2013 Aug 13. PMID 23794256
- [Result] Katzmarzyk PT, Mire E, Bray GA, Greenway FL, Heymsfield SB, Bouchard C. Anthropometric markers of obesity and mortality in white and African American adults: the pennington center longitudinal study. Obesity (Silver Spring). 2013 May;21(5):1070-5. doi: 10.1002/oby.20151. PMID 23784912
- [Result] Katzmarzyk PT, Hu G, Cefalu WT, Mire E, Bouchard C. The importance of waist circumference and BMI for mortality risk in diabetic adults. Diabetes Care. 2013 Oct;36(10):3128-30. doi: 10.2337/dc13-0219. Epub 2013 Jun 11. PMID 23757429
- [Result] Katzmarzyk PT, Heymsfield SB, Bouchard C. Clinical utility of visceral adipose tissue for the identification of cardiometabolic risk in white and African American adults. Am J Clin Nutr. 2013 Mar;97(3):480-6. doi: 10.3945/ajcn.112.047787. Epub 2013 Jan 30. PMID 23364010
- [Result] Katzmarzyk PT, Mire E, Bouchard C. Abdominal obesity and mortality: The Pennington Center Longitudinal Study. Nutr Diabetes. 2012 Aug 27;2(8):e42. doi: 10.1038/nutd.2012.15. PMID 23168527
- [Result] Camhi SM, Katzmarzyk PT. Total and femoral neck bone mineral density and physical activity in a sample of men and women. Appl Physiol Nutr Metab. 2012 Oct;37(5):947-54. doi: 10.1139/h2012-075. Epub 2012 Jul 23. PMID 22823076
- [Result] Barreira TV, Staiano AE, Harrington DM, Heymsfield SB, Smith SR, Bouchard C, Katzmarzyk PT. Anthropometric correlates of total body fat, abdominal adiposity, and cardiovascular disease risk factors in a biracial sample of men and women. Mayo Clin Proc. 2012 May;87(5):452-60. doi: 10.1016/j.mayocp.2011.12.017. PMID 22560524
- [Result] Barreira TV, Harrington DM, Staiano AE, Heymsfield SB, Katzmarzyk PT. Body adiposity index, body mass index, and body fat in white and black adults. JAMA. 2011 Aug 24;306(8):828-30. doi: 10.1001/jama.2011.1189. No abstract available. PMID 21862743
- [Result] Katzmarzyk PT, Barreira TV, Harrington DM, Staiano AE, Heymsfield SB, Gimble JM. Relationship between abdominal fat and bone mineral density in white and African American adults. Bone. 2012 Feb;50(2):576-9. doi: 10.1016/j.bone.2011.04.012. Epub 2011 Apr 28. PMID 21549867
- [Result] Hu G, Bouchard C, Bray GA, Greenway FL, Johnson WD, Newton RL Jr, Ravussin E, Ryan DH, Katzmarzyk PT. Trunk versus extremity adiposity and cardiometabolic risk factors in white and African American adults. Diabetes Care. 2011 Jun;34(6):1415-8. doi: 10.2337/dc10-2019. Epub 2011 Apr 19. PMID 21505210
- [Result] Katzmarzyk PT, Bray GA, Greenway FL, Johnson WD, Newton RL Jr, Ravussin E, Ryan DH, Bouchard C. Ethnic-specific BMI and waist circumference thresholds. Obesity (Silver Spring). 2011 Jun;19(6):1272-8. doi: 10.1038/oby.2010.319. Epub 2011 Jan 6. PMID 21212770
- [Result] Newton RL Jr, Bouchard C, Bray G, Greenway F, Johnson WD, Ravussin E, Ryan D, Katzmarzyk PT. Abdominal adiposity depots are correlates of adverse cardiometabolic risk factors in Caucasian and African-American adults. Nutr Diabetes. 2011 Jan 31;1(1):e2. doi: 10.1038/nutd.2010.2. PMID 23154294
- [Result] Broyles ST, Bouchard C, Bray GA, Greenway FL, Johnson WD, Newton RL, Ravussin E, Ryan DH, Smith SR, Katzmarzyk PT. Consistency of fat mass--fat-free mass relationship across ethnicity and sex groups. Br J Nutr. 2011 Apr;105(8):1272-6. doi: 10.1017/S0007114510004794. Epub 2010 Dec 14. PMID 21156087
- [Result] Sullivan R, Johnson WD, Katzmarzyk PT. Waist circumference is an independent correlate of errors in self-reported BMI. Obesity (Silver Spring). 2010 Nov;18(11):2237-9. doi: 10.1038/oby.2010.178. Epub 2010 Aug 19. PMID 20725063
- [Result] Katzmarzyk PT, Bray GA, Greenway FL, Johnson WD, Newton RL Jr, Ravussin E, Ryan DH, Smith SR, Bouchard C. Racial differences in abdominal depot-specific adiposity in white and African American adults. Am J Clin Nutr. 2010 Jan;91(1):7-15. doi: 10.3945/ajcn.2009.28136. Epub 2009 Oct 14. PMID 19828714
- [Result] Johnson WD, Bouchard C, Newton RL Jr, Ryan DH, Katzmarzyk PT. Ethnic differences in self-reported and measured obesity. Obesity (Silver Spring). 2009 Mar;17(3):571-7. doi: 10.1038/oby.2008.582. Epub 2008 Dec 18. PMID 19238143
- [Result] Camhi SM, Bray GA, Bouchard C, Greenway FL, Johnson WD, Newton RL, Ravussin E, Ryan DH, Smith SR, Katzmarzyk PT. The relationship of waist circumference and BMI to visceral, subcutaneous, and total body fat: sex and race differences. Obesity (Silver Spring). 2011 Feb;19(2):402-8. doi: 10.1038/oby.2010.248. Epub 2010 Oct 14. PMID 20948514
- [Result] Staiano AE, Bouchard C, Katzmarzyk PT. BMI-specific waist circumference thresholds to discriminate elevated cardiometabolic risk in White and African American adults. Obes Facts. 2013;6(4):317-24. doi: 10.1159/000354712. Epub 2013 Aug 9. PMID 23970141
- [Result] Sung YJ, Perusse L, Sarzynski MA, Fornage M, Sidney S, Sternfeld B, Rice T, Terry JG, Jacobs DR Jr, Katzmarzyk P, Curran JE, Jeffrey Carr J, Blangero J, Ghosh S, Despres JP, Rankinen T, Rao DC, Bouchard C. Genome-wide association studies suggest sex-specific loci associated with abdominal and visceral fat. Int J Obes (Lond). 2016 Apr;40(4):662-74. doi: 10.1038/ijo.2015.217. Epub 2015 Oct 20. PMID 26480920
- [Result] Katzmarzyk PT, Brown JC, Yang S, Mire EF, Wu XC, Miele L, Ochoa AC, Zabaleta J. Association of Abdominal Visceral Adiposity and Total Fat Mass with Cancer Incidence and Mortality in White and Black Adults. Cancer Epidemiol Biomarkers Prev. 2022 Aug 2;31(8):1532-1538. doi: 10.1158/1055-9965.EPI-22-0207. PMID 35654355
- [Result] Brown JC, Yang S, Mire EF, Wu X, Miele L, Ochoa A, Zabaleta J, Katzmarzyk PT. Obesity and cancer death in white and black adults: A prospective cohort study. Obesity (Silver Spring). 2021 Dec;29(12):2119-2125. doi: 10.1002/oby.23290. Epub 2021 Oct 24. PMID 34693655
- [Result] Brown JC, Yang S, Mire EF, Wu X, Miele L, Ochoa A, Zabaleta J, Katzmarzyk PT. Obesity and Cancer Risk in White and Black Adults: A Prospective Cohort Study. Obesity (Silver Spring). 2021 Jun;29(6):960-965. doi: 10.1002/oby.23163. PMID 34029447